CLINICAL TRIAL: NCT02222259
Title: A Feasibility Trial of Geriatric Assessment and Management for Older Cancer Patients (A GEM Study for Older Cancer Patients)
Brief Title: A Feasibility Trial of Geriatric Assessment and Management for Older Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Martine Puts, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14-7879-CE
Record Dates: First submitted 2014-08-18; First posted 2014-08-21 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer; Gastrointestinal Cancer; Genitourinary Cancer
Keywords: Geriatric Oncology; Quality of Life; Comprehensive Geriatric Assessment; Functional Status; Chemotherapy; Older Adults
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms; Urogenital Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GA and Integrated Care Plan (Experimental): Participants allocated to the intervention group will be seen in the geriatric oncology clinic where they will be assessed using a geriatric assessment. Based on the issues identified in the geriatric assessment, a care plan will be developed with the participant to address the issues.
  Interventions: Procedure: GA and Integrated Care Plan
- Standard oncology care (No Intervention): Participants randomized to standard oncology care will receive usual care from their oncology team.

INTERVENTIONS:
Procedure: GA and Integrated Care Plan — The intervention will consist of a Geriatric Assessment conducted by a multidisciplinary geriatric oncology team followed by an integrated care plan developed and implemented by the team for those issues identified in the assessment. The study intervention includes contact with the intervention team at 4 points in time during the study: at baseline (to conduct the assessment and develop the integrated care plan), 2-3 weeks by telephone after the clinic visit to evaluate if the plan needs adjustments, at 3 and 6 months (to evaluate the outcomes of the integrated care plan; i.e., did the patient follow all recommendations of the integrated care plan and did the plan lead to the desired outcomes for the problems identified?
  Arms: GA and Integrated Care Plan

SUMMARY:
The purpose of this study is to determine the feasibility of implementing a randomized controlled study of the intervention (Geriatric Assessment followed by an integrated care plan carried out by the multidisciplinary geriatric oncology team) designed to maintain/improve quality of life and functional status in older adults with advanced gastrointestinal, genitourinary or breast cancer referred for first line chemotherapy.

Secondarily, the study will investigate the impact of the Geriatric Assessment on the cancer treatment decision of the cancer specialist.

DETAILED DESCRIPTION:
Introduction: A comprehensive geriatric assessment (CGA) can identify functional and psychosocial issues in older cancer patients, which in turn can inform interventions to prevent/postpone adverse outcomes and maintain/improve the functional status and well-being of this population. However, few randomized controlled trials (RCTs) have been completed showing the evidence.

OBJECTIVE - To explore the feasibility and impact of a CGA followed by an integrated care plan on quality of life and functional status for older adults with advanced breast, gastrointestinal or genitourinary cancer METHODS -

A two-group parallel single-blind phase II RCT is enrolling 60 patients aged 70 or above, diagnosed with cancer, and starting first line chemotherapy at Princess Margaret Cancer Centre in Toronto. The randomization using sealed opaque envelopes is stratified by treatment intent (adjuvant versus palliative). The intervention entails a comprehensive CGA by a multidisciplinary geriatric oncology team followed by an integrated care plan to address any issues identified. Participants in the intervention group are seen at baseline for the CGA and for initiation of the integrated care plan, and again at 3 and 6 months to assess intervention fidelity and measure outcomes. The co-primary outcomes are: 1) maintaining/improvement in quality of life; 2) refining of cancer treatment plan. The secondary outcomes include: 1) Functional status; 2) feasibility of the study by tumor site.

Recruitment has been completed November 2015

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of advanced (stage 2, 3 or 4) Gastrointestinal, Genitourinary, or breast cancer
* Referred for first-line chemotherapy
* Ability to speak English
* Physician estimated life expectancy >6 months
* An Eastern Oncology Group Collaborative (ECOG) Performance Score of 0-2
* Ability to provide informed consent

Exclusion Criteria:

* Previous chemotherapy for current stage of disease

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Quality of life | 6 months
  We will measure quality of life with European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core version 30 items (EORTC QLQ C30)

SECONDARY OUTCOMES:
Impact of the Geriatric Assessment (GA) on the cancer treatment decision questionnaire | 6 months
  The treating oncologist will be asked to indicate the cancer treatment plan prior to receiving the geriatric assessment results using a survey previously used in the study of Dr. Alibhai et al (Am J Clin Oncol. 2012 Aug;35(4):322-8.).
  After the GA the results will be send to the treating oncologist and after the physician will be asked to indicate whether or not and if yes how he/she modified the treatment plan based on the GA results
Functional status | 6 months
  We will measure functional status with the Older American Resources and Services Instrumental Activities of Daily Living questionnaire (7 items)

CONTACTS AND LOCATIONS:
Overall Officials: Shabbir Alibhai, MD, Principal Investigator — University Health Network, Toronto; Martine Puts, PhD, Principal Investigator — University of Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Sattar S, Alibhai SMH, Brennenstuhl S, Kulik M, MacDonald ME, McWatters K, Lee K, Jang R, Amir E, Krzyzanowska MK, Joshua AM, Monette J, Wan-Chow-Wah D, Puts MTE. Health status, emergency department visits, and oncologists' feedback: An analysis of secondary endpoints from a randomized phase II geriatric assessment trial. J Geriatr Oncol. 2019 Jan;10(1):169-174. doi: 10.1016/j.jgo.2018.06.014. Epub 2018 Jul 21. PMID 30041978
- [Derived] Puts MTE, Sattar S, Kulik M, MacDonald ME, McWatters K, Lee K, Brennenstuhl S, Jang R, Amir E, Krzyzanowska MK, Joshua AM, Monette J, Wan-Chow-Wah D, Alibhai SMH. A randomized phase II trial of geriatric assessment and management for older cancer patients. Support Care Cancer. 2018 Jan;26(1):109-117. doi: 10.1007/s00520-017-3820-7. Epub 2017 Jul 25. PMID 28741175